CLINICAL TRIAL: NCT06443047
Title: Suturing Through-the-scope System Used for Prophylactic Closure of Colonic Post-ESD Defects: A Randomized Trial vs Conventional Clips That it Highlights the Importance of Suturing in Promoting Healing and Closure of the Colonic ESD Defects
Brief Title: Suturing Through-the-scope System Used for Prophylactic Closure of Colonic Post-ESD Defects
Acronym: STITCH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3938 - STITCH
Record Dates: First submitted 2024-05-24; First posted 2024-06-05 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Precancerous Lesion of Colon
Keywords: precancerous colorectal lesions

STUDY DESIGN:
Intervention Model Description: The goal of this study is to perform a randomized trial to compare a new through-the-scope suturing system and conventional clips for closure of defect after ESD for 30-60 mm colonic polyps. More precisely, the hypothesis posits that the new through-the-scope suturing system can achieve higher complete closure rates in a shorter time in comparison to conventional clips.
  Considering an α risk set at 5%, a power set at 80%, given an expected complete resection rate of 70% in the control group and of 95% in the experimental group, 33 patients in each group are required. Thus, the investigators will enroll 66 subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ESD with clips (No Intervention): Closure of the defect will be performed at the end of the Endoscopic Submucosal Dissection procedure with clips (Boston scientific®). Pictures or movies of the closing defect will be necessary to independently confirm the complete closure.
- TTS suturing system (Experimental): Closure of the defect will be performed at the end of the ESD procedure with a new TTS suturing system (X-Tack Boston scientific®). Pictures or movies of the closing defect will be necessary to independently confirm the complete closure.
  Interventions: Device: TTS suturing system

INTERVENTIONS:
Device: TTS suturing system — The use of TTS suturing system could allow a quick, complete endoscopic closure of colonic post-ESD defects, providing relevant clinical and medico-economic benefits.
  Arms: TTS suturing system

SUMMARY:
The goal of this study is to perform a randomized trial to compare a new through-the-scope suturing system and conventional clips for closure of defect after ESD for 30-60 mm colonic polyps. More precisely, the hypothesis posits that the new through-the-scope suturing system can achieve higher complete closure rates in a shorter time in comparison to conventional clips.

DETAILED DESCRIPTION:
Large superficial colonic polyps are increasingly detected thanks to colorectal cancer screening programs worldwide. ESD is the technique which provides a high-quality resection of these large polyps.

Nevertheless, several adverse events affect ESD, especially in the colon. They could be life-threatening, call for or prolong the hospitalization, require blood transfusion, additional endoscopic or surgical procedures and increase costs.

Thus, preventing these adverse events is an important clinical and medico-economic objective. Endoscopic closure of post-ESD defects could reduce this risk. However, closing these large defects with conventional clips can be difficult, unsuccessful and prolong the duration of the whole procedure. A new trough-the-scope suturing system could successfully provide a complete endoscopic closure of post-ESD defects in the colon in a reasonable time.

Expected benefits are a decrease of morbidity and costs related to colonic ESD procedure

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from 30-60 mm colonic polyps with indication of ESD
* Male or female patients aged > 18 years' old
* Patients able to fill in questionnaires written in Italian

Exclusion Criteria:

* Failure of endoscopic resection
* Suspicion of deep submucosal cancer by analysis of pit pattern (KUDO Vn)
* Polyp involving the appendix deeply (type 2 or 3 according to Toyonaga classification)
* Polyp inside the ileo-cecal valvula.
* Rectal lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Compare the proportion of complete closure between the two groups | Intra-procedural
  To assess the proportion of complete closure, defined when opposite margins are drawn together without a persistent post-resection defect of more than 1 cm (pictures and/or videos)

SECONDARY OUTCOMES:
duration of the closure procedure | up to 2 hours
  To assess the closure procedure time, which is defined by duration between the beginning of assemblage of the suturing system and the end of the closure in the intervention group and between the opening of the bag of the first clip until the end of the closure in the control group.(pictures-videos)

OTHER OUTCOMES:
Proportion of post-polypectomy syndrome | 1 week
  To assess, it will compare the proportion between the 2 groups of post-polypectomy syndrome at Day 7
Proportion of clinically significant delayed bleeding | 1 month
  Compare and assess the proportion of clinically significant delayed bleeding at 1 month
Cost-effectiveness ratio | 1 month
  To assess the cost-effectiveness ratio, estimated by dividing the difference in costs observed between the two strategies by the difference of effectiveness at 1 month. The effectiveness criterion being the closure time at 1 month
Length of hospitalization | up to 1 week
  To compare the length of hospitalization defined as the number of procedural nights in the hospitals

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Repici, Prof., Principal Investigator — IRCCS Humanitas Research Hospital - Rozzano 20089, Milan, Italy

REFERENCES:
- [Background] Morgan E, Arnold M, Gini A, Lorenzoni V, Cabasag CJ, Laversanne M, Vignat J, Ferlay J, Murphy N, Bray F. Global burden of colorectal cancer in 2020 and 2040: incidence and mortality estimates from GLOBOCAN. Gut. 2023 Feb;72(2):338-344. doi: 10.1136/gutjnl-2022-327736. Epub 2022 Sep 8. PMID 36604116
- [Background] Arnold M, Sierra MS, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global patterns and trends in colorectal cancer incidence and mortality. Gut. 2017 Apr;66(4):683-691. doi: 10.1136/gutjnl-2015-310912. Epub 2016 Jan 27. PMID 26818619
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2018. CA Cancer J Clin. 2018 Jan;68(1):7-30. doi: 10.3322/caac.21442. Epub 2018 Jan 4. PMID 29313949
- [Background] Schoen RE, Pinsky PF, Weissfeld JL, Yokochi LA, Church T, Laiyemo AO, Bresalier R, Andriole GL, Buys SS, Crawford ED, Fouad MN, Isaacs C, Johnson CC, Reding DJ, O'Brien B, Carrick DM, Wright P, Riley TL, Purdue MP, Izmirlian G, Kramer BS, Miller AB, Gohagan JK, Prorok PC, Berg CD; PLCO Project Team. Colorectal-cancer incidence and mortality with screening flexible sigmoidoscopy. N Engl J Med. 2012 Jun 21;366(25):2345-57. doi: 10.1056/NEJMoa1114635. Epub 2012 May 21. PMID 22612596
- [Background] Nishihara R, Wu K, Lochhead P, Morikawa T, Liao X, Qian ZR, Inamura K, Kim SA, Kuchiba A, Yamauchi M, Imamura Y, Willett WC, Rosner BA, Fuchs CS, Giovannucci E, Ogino S, Chan AT. Long-term colorectal-cancer incidence and mortality after lower endoscopy. N Engl J Med. 2013 Sep 19;369(12):1095-105. doi: 10.1056/NEJMoa1301969. PMID 24047059
- [Background] Jacques J, Schaefer M, Wallenhorst T, Rosch T, Lepilliez V, Chaussade S, Rivory J, Legros R, Chevaux JB, Leblanc S, Rostain F, Barret M, Albouys J, Belle A, Labrunie A, Preux PM, Lepetit H, Dahan M, Ponchon T, Crepin S, Marais L, Magne J, Pioche M. Endoscopic En Bloc Versus Piecemeal Resection of Large Nonpedunculated Colonic Adenomas : A Randomized Comparative Trial. Ann Intern Med. 2024 Jan;177(1):29-38. doi: 10.7326/M23-1812. Epub 2023 Dec 12. PMID 38079634
- [Background] Arezzo A, Passera R, Marchese N, Galloro G, Manta R, Cirocchi R. Systematic review and meta-analysis of endoscopic submucosal dissection vs endoscopic mucosal resection for colorectal lesions. United European Gastroenterol J. 2016 Feb;4(1):18-29. doi: 10.1177/2050640615585470. Epub 2015 May 5. PMID 26966519
- [Background] Liu M, Zhang Y, Wang Y, Zhu H, Xu H. Effect of prophylactic closure on adverse events after colorectal endoscopic submucosal dissection: A meta-analysis. J Gastroenterol Hepatol. 2020 Nov;35(11):1869-1877. doi: 10.1111/jgh.15148. Epub 2020 Jul 5. PMID 32542857
- [Background] Dong L, Zhu W, Zhang X, Xie X. Does Prophylactic Closure Improve Outcomes After Colorectal Endoscopic Submucosal Dissection? A Systematic Review and Meta-analysis. Surg Laparosc Endosc Percutan Tech. 2024 Feb 1;34(1):94-100. doi: 10.1097/SLE.0000000000001248. PMID 38011072
- [Background] Pohl H, Grimm IS, Moyer MT, Hasan MK, Pleskow D, Elmunzer BJ, Khashab MA, Sanaei O, Al-Kawas FH, Gordon SR, Mathew A, Levenick JM, Aslanian HR, Antaki F, von Renteln D, Crockett SD, Rastogi A, Gill JA, Law RJ, Elias PA, Pellise M, Wallace MB, Mackenzie TA, Rex DK. Clip Closure Prevents Bleeding After Endoscopic Resection of Large Colon Polyps in a Randomized Trial. Gastroenterology. 2019 Oct;157(4):977-984.e3. doi: 10.1053/j.gastro.2019.03.019. Epub 2019 Mar 15. PMID 30885778
- [Background] Kobara H, Tada N, Fujihara S, Nishiyama N, Masaki T. Clinical and technical outcomes of endoscopic closure of postendoscopic submucosal dissection defects: Literature review over one decade. Dig Endosc. 2023 Jan;35(2):216-231. doi: 10.1111/den.14397. Epub 2022 Aug 25. PMID 35778927
- [Background] Farha J, Ramberan H, Aihara H, Zhang LY, Mehta A, Hage C, Schlachterman A, Kumar A, Shinn B, Canakis A, Kim RE, D'Souza LS, Buscaglia JM, Storm AC, Samarasena J, Chang K, Friedland S, Draganov PV, Qumseya BJ, Jawaid S, Othman MO, Hasan MK, Yang D, Khashab MA, Ngamruengphong S; ESD-Closure working group. A novel through-the-scope helix tack-and-suture device for mucosal defect closure following colorectal endoscopic submucosal dissection: a multicenter study. Endoscopy. 2023 Jun;55(6):571-577. doi: 10.1055/a-1970-5528. Epub 2022 Nov 2. PMID 36323330